CLINICAL TRIAL: NCT02552355
Title: Milk Protein Feeding After Aerobic Exercise in Older Adults With Pre-diabetes Taking the Biguanide Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Benjamin Miller, Associate Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-8573H
Record Dates: First submitted 2015-09-01; First posted 2015-09-17 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either Metformin-Protein, Metformin-Carbohydrate, Placebo-Protein, and Placebo-Carbohydrate.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metformin/Carbohydrate (Experimental): Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. The dose of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4. Supervised aerobic exercise 3 days per week followed by a carbohydrate drink along with daily oral administration of Metformin.
  Interventions: Drug: Metformin; Dietary Supplement: Carbohydrate Beverage
- Placebo/Carbohydrate (Placebo Comparator): Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4. Supervised aerobic exercise 3 days per week followed by a carbohydrate drink along with daily oral administration of matching placebo.
  Interventions: Drug: Placebo; Dietary Supplement: Carbohydrate Beverage
- Metformin/Protein (Active Comparator): Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. The dose of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week. Supervised aerobic exercise 3 days per week followed by a protein drink along with daily oral administration of Metformin
  Interventions: Drug: Metformin; Dietary Supplement: Protein Beverage
- Placebo/Protein (Active Comparator): Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. The dose of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week. Supervised aerobic exercise 3 days per week followed by a protein drink along with daily oral administration of placebo.
  Interventions: Drug: Placebo; Dietary Supplement: Protein Beverage

INTERVENTIONS:
Drug: Metformin — Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
  Other Names: Glumetza; Fortamet; Glucophage; Riomet
  Arms: Metformin/Carbohydrate; Metformin/Protein
Drug: Placebo — Daily administration of matching placebo during a 12 week exercise training program.
  Arms: Placebo/Carbohydrate; Placebo/Protein
Dietary Supplement: Carbohydrate Beverage — Supervised aerobic exercise 3 days per week followed by a carbohydrate drink
  Arms: Metformin/Carbohydrate; Placebo/Carbohydrate
Dietary Supplement: Protein Beverage — Supervised aerobic exercise 3 days per week followed by a protein drink
  Arms: Metformin/Protein; Placebo/Protein

SUMMARY:
The investigators propose that post-exercise milk protein feeding will enhance the mitochondrial protein synthesis (biogenesis) response to an exercise-training program. In addition, the investigators propose that this stimulatory effect of protein feeding will overcome the potential blunting effect of metformin on exercise responses. The investigators will investigate these outcomes over a 12-week exercise-training program in older adults with pre-diabetes with or without metformin treatment.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double blind study. 60 men and women over the age of 55 with indications of pre-diabetes will be recruited for participation and randomly assigned to one of four 12 week exercise training programs: 1)Supervised aerobic exercise 3 days per week followed by a carbohydrate drink along with daily oral administration of Metformin. 2) Supervised aerobic exercise 3 days per week followed by a protein drink along with daily oral administration of Metformin. 3) Supervised aerobic exercise 3 days per week followed by a carbohydrate drink along with daily oral administration of matching placebo. 4) Supervised aerobic exercise 3 days per week followed by a protein drink along with daily oral administration of placebo.

Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program. The titration dosing scheme and taking metformin/placebo with meals will help reduce the most common side effects (i.e.,gastrointestinal discomfort). If participants experience gastrointestinal discomfort, the dose will be lowered to 1500 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Individuals with Prediabetes defined as impaired fasting glucose (100 to 126 mg/dl), HbA1c (5.7-6.4%), and/or impaired glucose tolerance defined as 2 hour postprandial blood glucose of 140 to 200 mg/dl.

Exclusion Criteria:

* Medications contraindicated with Metformin (Dofetilide, Lamotrigine, Pegvisomant, Somatropin, Trimethoprim, Trospium, Gatifloxacin, Cephalexin, Cimetidine, Dalfampridine)
* Recent (less than 6 weeks) or planned imaging that requires IV contrast,
* Renal dysfunction creatinine ≥ 1.3 mg/dL in men or ≥ 1.2 mg/dL in women
* Alanine Aminotransferase (ALT) levels exceed 52 IU/L
* Heart, Kidney or Liver Disease
* Type I or Type II Diabetes
* Anti-coagulant therapy (warfarin/heparin)
* Lung/respiratory dysfunction
* Medications affecting primary outcomes
* Lactose Intolerant
* Tobacco Use
* Heavy Alcohol Use
* Cancer
* Lidocaine Allergy

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

REFERENCES:
- See also: Lab website — http://tracd.colostate.edu/
- See also: Final Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6351883/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to either Metformin-Protein, Metformin-Carbohydrate, Placebo-Protein, and Placebo-Carbohydrate.
Groups:
- Metformin:Carbohydrate: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a isocaloric carbohydrate beverage.
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo:Carbohydrate: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of with post-exercise consumption of a protein beverage. The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Placebo: Daily administration of matching placebo during a 12 week exercise training program.
- Metformin:Protein: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a protein beverage. The dose of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4.
- Placebo: Carbohydrate: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a isocaloric carbohydrate beverage. The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
Period: Overall Study
Arm/Group | Metformin:Carbohydrate | Placebo:Carbohydrate | Metformin:Protein | Placebo: Carbohydrate
Started | 14 | 13 | 14 | 15
Completed | 14 | 11 | 12 | 14
Not Completed | 0 | 2 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 subjects were withdrawn from the Placebo: Carbohydrate group (1 subject's baseline data was analyzed). 2 subjects were withdrawn from the Metformin: Protein group (1 subject's baseline data was analyzed). 1 subject was withdrawn from the Placebo: Protein Group and baseline data was not analyzed.
Groups:
- Metformin: Carbohydrate: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. Immediately after each exercise session, participants consumed a standardized beverage that consisted of carbohydrates (82g) plus protein (2g).
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo: Carbohydrate: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Immediately after each exercise session, participants consumed a standardized beverage that consisted of carbohydrates (82g) plus protein (2g).
- Metformin: Protein: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training. Immediately after each exercise session, participants consumed a standardized beverage that consisted of carbohydrate (63g) plus protein (20g).
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo: Protein: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Immediately after each exercise session, participants consumed a standardized beverage that consisted of carbohydrates (63 g) plus protein (20g).
- Total: Total of all reporting groups
Arm/Group | Metformin: Carbohydrate | Placebo: Carbohydrate | Metformin: Protein | Placebo: Protein | Total
Number analyzed (Participants) | 14 | 12 | 13 | 14 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 13 | 14 | 53
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 10 | 11 | 42
  Male | 3 | 2 | 3 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 14 | 12 | 13 | 14 | 53
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 13 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Mitochondrial Function
Description: Oxygen consumption was assessed via high-resolution mitochondrial respirometry in permeabilized skeletal muscle. This outcome was assessed via 2 different protocols; Protocol 1 was a substrate-uncoupler-inhibitor titration (SUIT) and Protocol 2 was an adenosine diphosphate (ADP) titration. These data are reported as the percent change from baseline compared to 12 weeks.
Time Frame: Baseline and 12 weeks
Population: The number analyzed differs from the overall number due to subject withdrawal from study and/or limited muscle sample.
Measure: Mean (Standard Error); unit: percent change in pmol/s/mg tissue
Groups:
- Metformin: Carbohydrate: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a carbohydrate beverage.
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo:Carbohydrate: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Placebo: Daily administration of matching placebo during a 12 week exercise training program with post-exercise consumption of a carbohydrate beverage.
- Metformin: Protein: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a protein beverage.
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo: Protein: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Placebo: Daily administration of matching placebo during a 12 week exercise training program with post-exercise consumption of a protein beverage.
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 13 | 14
percent change in pmol/s/mg tissue
  SUIT: number analyzed (Participants) | 14 | 11 | 13 | 14
  SUIT | 7.1 (12.8) | 43.2 (15.5) | 15.6 (7.6) | 13.8 (6.9)
  ADP titration: number analyzed (Participants) | 14 | 11 | 13 | 14
  ADP titration | 3.4 (8.2) | 42.3 (12.9) | 4.7 (11.7) | 16 (9.4)

2. Primary Outcome: Protein Synthesis
Description: Incorporation of deuterium into proteins to calculate cumulative synthesis rates. Protein synthesis was measured in sub cellular fractions of skeletal muscle including mixed, cytoplasmic and mitochondrial enriched fractions. These data are reported as the mean at 12 weeks.
Time Frame: 12 weeks
Population: The number analyzed differs from the over all number due to subject withdrawal from study and/or limited muscle sample.
Measure: Mean (Standard Error); unit: % of protein synthesis rate per day
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 12 | 14
% of protein synthesis rate per day
  Mixed: number analyzed (Participants) | 13 | 11 | 11 | 14
  Mixed | 1.24 (0.06) | 1.15 (0.04) | 1.1 (0.04) | 1.14 (0.04)
  Cytoplasmic: number analyzed (Participants) | 14 | 11 | 11 | 14
  Cytoplasmic | 1.15 (0.07) | 1.00 (0.05) | 1.05 (0.03) | 1.06 (0.05)
  Mitochondrial: number analyzed (Participants) | 13 | 12 | 12 | 14
  Mitochondrial | 1.09 (0.09) | 0.97 (0.08) | 1.03 (0.04) | 0.95 (0.07)

3. Primary Outcome: Body Composition
Description: Dual energy x-ray absorptiometry was used to assess fat-free and fat mass. These data are reported as the mean at baseline (pre) and mean at 12 weeks (post).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 13 | 14
Kilograms
  Pre Fat Free Mass | 48 (3) | 48 (3) | 50 (2) | 46 (2)
  Post Fat Free Mass | 47 (2) | 48 (2) | 50 (3) | 46 (2)
  Pre Fat Mass | 34 (3) | 35 (3) | 33 (3) | 33 (4)
  Post Fat Mass | 32 (3) | 34 (2) | 31 (3) | 32 (4)

4. Primary Outcome: Insulin Sensitivity
Description: Oral glucose tolerance test was used to measure whole-body insulin sensitivity. These data are reported as the mean at baseline (pre) and the mean at 12 weeks (post).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: microInternational units/mL
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 13 | 14
microInternational units/mL
  Pre 2 hour Insulin | 86 (20) | 57 (14) | 39 (7) | 56 (13)
  Post 2 hour Insulin | 91 (34) | 51 (8) | 32 (7) | 55 (15)

5. Primary Outcome: Peak Aerobic Capacity
Description: Indirect calorimetry was used to measure peak oxygen consumption during a maximal, graded exercise test. These data are reported as the percent change from baseline compared to 12 weeks.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percent change of Liters/Minute
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 13 | 13
percent change of Liters/Minute | 3 (2.1) | 4.7 (3.8) | 4.9 (2.8) | 8.5 (2.9)

6. Primary Outcome: DNA Synthesis
Description: Incorporation of Deuterium Oxide into DNA will be measured before and after the 12 week interventions.
Time Frame: Baseline and 12 weeks
Population: No data was collected.
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Intracellular Signaling Proteins
Description: Protein content of intracellular signaling proteins that are implicated in mitochondrial biogenesis, mitochondrial function and insulin sensitivity were measured by Western blotting. Densitometry results are reported as a ratio of protein divided by total amount of protein expressed. All proteins of interest are expressed as phosphorylated relative to total. These data are reported as the percent change from baseline compared to 12 weeks.
Time Frame: Baseline and 12 weeks
Population: Proteins were analyzed in a subset of participants due to limited tissue availability.
Measure: Mean (Standard Error); unit: percent change of densitometry ratio
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 10 | 8 | 13
percent change of densitometry ratio
  Ratio of AKT S473 phospho/total): number analyzed (Participants) | 9 | 8 | 7 | 10
  Ratio of AKT S473 phospho/total) | 154.3 (46.7) | 677.5 (187.5) | 321.1 (147.4) | 106.9 (28.8)
  ratio of AKT T308 phospho /total): number analyzed (Participants) | 9 | 8 | 7 | 10
  ratio of AKT T308 phospho /total) | 151.8 (43.2) | 563.2 (230.1) | 477.3 (148.2) | 94.0 (25.4)
  RPS6 ratio of phospho/total: number analyzed (Participants) | 14 | 10 | 7 | 13
  RPS6 ratio of phospho/total | 16.6 (12.6) | -2.2 (25.4) | 47.0 (16.5) | -15.6 (15.4)
  4EBP1 ratio of phospho/total: number analyzed (Participants) | 14 | 8 | 8 | 12
  4EBP1 ratio of phospho/total | 35 (25.2) | 57 (42) | 122 (76) | 13.5 (13.9)

8. Secondary Outcome: Glucose Profiles From Real-Time Continuous Glucose Monitoring
Description: Data derived from Continuous Glucose Monitoring was used to calculate mean glucose and mean average glucose excursions (MAGE). These data are reported as the percent change at baseline (pre), 6-8 weeks (Mid), and 12 weeks (post) .
Time Frame: Baseline, Weeks 6-8, 12 weeks
Population: Only a subset of subjects were studied.
Measure: Mean (Standard Error); unit: percent change of milligrams/deciliter
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 4 | 4 | 4 | 5
percent change of milligrams/deciliter
  Mean Glucose- Pre | 116 (9.9) | 116.7 (5.9) | 113.3 (3.5) | 107.1 (5.3)
  Mean Glucose- Mid | 105.3 (6.2) | 104.7 (4.1) | 93.7 (7.7) | 95.2 (10.7)
  Mean Glucose-Post | 110.7 (2.7) | 116.1 (6.2) | 107.8 (3.7) | 108.6 (2.0)
  MAGE- Pre | 61.3 (15) | 49.5 (4.2) | 41.1 (3.0) | 46.4 (6.5)
  MAGE- Mid | 53.6 (6.9) | 40.8 (3.1) | 36.2 (2.5) | 37.1 (4.9)
  MAGE- Post | 56.4 (8.4) | 58.6 (7.1) | 42.1 (2.9) | 46.3 (5.5)

9. Primary Outcome: Glucose Tolerance
Description: Oral glucose tolerance test was used to measure glucose tolerance. These data are reported as the mean at baseline (pre) and the mean at 12 weeks (post).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin: Carbohydrate | Placebo:Carbohydrate | Metformin: Protein | Placebo: Protein
Number analyzed (Participants) | 14 | 12 | 13 | 14
mg/dL
  Pre 2 hour Glucose | 131 (7) | 116 (7) | 108 (14) | 102 (7)
  Post 2 hour Glucose | 133 (7) | 115 (7) | 112 (12) | 107 (10)

ADVERSE EVENTS:
Time Frame: From the start of the intervention period through the 12 week intervention period.
Description: Participants were assigned to either Metformin-Protein, Metformin-Carbohydrate, Placebo-Protein, and Placebo-Carbohydrate.
Groups:
- Metformin: Carbohydrate: Daily oral administration of Metformin with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training with post-exercise consumption of a isocaloric carbohydrate beverage.
  Metformin: Daily administration of Metformin will begin as one 500 mg tablet for the first week and will increase by 500 mg/day/week until reaching 2000 mg/day by week 4 during a 12 week exercise training program.
- Placebo: Carbohydrate: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Placebo: Daily administration of matching placebo during a 12 week exercise training program with post-exercise consumption of an isocaloric carbohydrate beverage.
- Placebo:Protein: Daily oral administration of matching placebo with a 12-week exercise training program consisting of 3 days per week of aerobic exercise training The dose of matching placebo will begin as one tablet for the first week and will increase by one tablet/day/week until reaching 4 tablets by week 4.
  Placebo: Daily administration of matching placebo during a 12 week exercise training program with post-exercise consumption of a protein beverage.
Arm/Group | Metformin: Carbohydrate | Placebo: Carbohydrate | Metformin: Protein | Placebo:Protein
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 5/14 | 5/13 | 9/14 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin: Carbohydrate (N=14) | Placebo: Carbohydrate (N=13) | Metformin: Protein (N=14) | Placebo:Protein (N=15)
Diarrhea/Nausea/Stomach Cramps (General disorders) | 5 (12) | 2 (2) | 5 (5) | 6 (8)
Leg Cramps/Muscle Soreness (General disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
High blood Pressure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
High Creatine (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Infection/Pressure (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hair Loss (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Common Cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headaches/Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02552355/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02552355/ICF_001.pdf